CLINICAL TRIAL: NCT02394678
Title: Rheolytic Thrombectomy For Adult Intraventricular Haemorrhage
Acronym: rtIVH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karol Palwel Budohoski (Other)
Responsible Party: Sponsor-Investigator, Karol Palwel Budohoski, Academic Clinical Fellow, Neurosurgery, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A093205
Record Dates: First submitted 2015-03-12; First posted 2015-03-20 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Intraventricular Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention - clot removal (Experimental): Patients will undergo rheolytic thrombectomy for intraventricular hemorrhage
  Interventions: Device: AngioJet Thrombectomy System

INTERVENTIONS:
Device: AngioJet Thrombectomy System — Mechanical removal of blood, using a pressurised jet of water, from ventricles of patients suffering from intraventricular haemorrhage

SUMMARY:
Intraventricular haemorrhage (IVH) - bleeding into the normal fluid spaces (ventricles) within the brain - is associated with a high risk of death or significant long-term disability. IVH leads to an increase pressure within the head and triggers inflammation and swelling in the surrounding brain. The ideal treatment for IVH would both rapidly relieve pressure and safely remove as much blood as possible to prevent any further injury to the brain. Currently, patients are managed by inserting a tube into the ventricle that drains fluid to the outside and helps reduce pressure, but does not address the blood clot itself, which naturally dissolves only over several days or weeks.

Furthermore, these drains frequently block because of blood clots that for within them. If that occurs a repeat operation is required to replace them. Experimental treatments include infusing drugs to accelerate clot breakdown but this can nonetheless still take a number of days and the process introduces a risk of infection and fresh bleeding. Surgery to remove the blood clot is hazardous, technically challenging, and generally not very successful. Therefore, at the present time, none of the available options achieve all the stated goals of IVH treatment and there is an unmet need for better interventions.

In this study the investigators propose to pilot a novel instrument that employs a high pressure but very localised microjet of water to mechanically disrupt blood clots and then sucks the debris away. This technique has been highly successful in reopening blocked arteries in the heart and, importantly, does so without damaging the underlying vessel lining. In the context of IVH, this should allow rapid removal of blood from the ventricles while causing minimal trauma to the brain. Clearing the blood early will prevent the build-up of pressure and inflammation, and improve the chances of patients making a good recovery.

DETAILED DESCRIPTION:
Intraventricular Haemorrhage Approximately 30% of cases of spontaneous intracranial haemorrhage or severe head injury are complicated by intraventricular haemorrhage (IVH). Typically, IVH results from extension of deep intracerebral haemorrhage (ICH) or aneurysmal subarachnoid haemorrhage (SAH), though a third of patients may have primary IVH confined solely the ventricular system. In the absence of a demonstrable angiographic abnormality IVH is usually associated with deranged coagulation or vascular risk factors such as hypertension, diabetes, and smoking.

Both experimental and clinical studies have clearly demonstrated the independent effect of the volume of haemorrhage on death and disability from IVH. In animals, injection of blood into the lateral ventricle exhibits a dose-dependent increase in the risk of fatality, and early thrombolysis of the simulated IVH reduces the severity of neurological deficit. In retrospective reports of intracerebral haemorrhage patient series concomitant IVH consistently emerges as a risk factor for greater mortality and poor functional outcome. Similarly, multivariate analyses of data from the STICH and FAST prospective randomised controlled trials of ICH management has provided conclusive evidence that the presence and volume of IVH is a significant independent risk factor for mortality and morbidity.

The principal effects of IVH are mediated by intracranial hypertension and induction of inflammation with oedema in the periventricular white matter and deep grey structures. Blood within the ventricles blocks CSF pathways resulting in a sequence of hydrocephalus, acute rise in intracranial pressure (ICP), reduced cerebral perfusion, with a risk of ischaemia, and potential brainstem herniation. Exposure of the ependymal lining to blood initiates inflammatory cascades and leucocyte infiltration into the adjacent brain, with ensuing tissue injury, localised oedema, and eventually generalised brain swelling. Late effects of IVH include scarring of the ventricles and obstruction of CSF absorption by blood breakdown products, typically resulting in chronic hydrocephalus necessitating permanent CSF diversion (shunting).

Current Management of Intraventricular Haemorrhage The rapid onset of deleterious effects after IVH supports the rationale of early intervention to relieve hydrocephalus and raised ICP, and to reduce blood load and the resulting inflammation and oedema. In most neurosurgical centres the prevailing treatment paradigm is insertion of a ventricular catheter and external drainage to divert CSF and reduce ICP, though this can be of limited efficacy with a large IVH as expansion and distortion of the ventricle by haematoma plays a greater role in exerting mechanical pressure than obstructed CSF. Ventricular catheters also frequently block with blood, necessitating repeated surgery for replacement. Furthermore, this mode of treatment does not address the inflammatory effects of the haematoma itself, which may persist for several days or weeks before complete reabsorption occurs. Infusions of urokinase or recombinant tissue plasminogen activator via an external drain to accelerate clot lysis have shown promise, however, the effect is not immediate and serial treatments are required, each with an attendant risk of infection and rebleeding. Several authors have described transcortical or endoscopic surgical clot evacuation but such approaches are technically demanding, have limited success in terms of the volume of haematoma removed, and are not practicable in the emergency situation.

Rheolytic Thrombectomy Rheolytic thrombectomy (RT) involves a double-lumen endovascular catheter that delivers multiple high-speed retrograde water jets to create a hydrodynamic recirculation vortex that traps and mechanically fragments adjacent thrombus, with the resulting debris evacuated via the continuous aspiration lumen. Safety studies have shown that the technique causes minimal denuding of vascular endothelium with no difference in the degree of vessel injury compared with traditional balloon thrombectomy. Clinically, RT has principally been applied to endovascular extraction of acute thrombus in coronary arteries and the results of large randomised controlled trials testify to a favourable safety profile. RT has also been used successfully to treat intracranial dural sinus thrombosis, acute internal carotid artery occlusion, and for recanalising blocked synthetic vascular grafts.

These attractive features of RT suggest it may offer significant advantages over conventional IVH treatment for rapidly removing clot from within the ventricle in a single procedure, while at the same time causing minimal trauma to the ependymal lining and brain. This study will evaluate the feasibility, safety, and efficacy of RT therapy for adult IVH.

Rationale There is an unmet need for interventions directed at early clot removal following IVH. RT has proven effective and safe for intravascular thrombectomy and its features suggest it has the potential to be similarly successful in the treatment of IVH. A pilot study is indicated to establish feasibility and safety as a precursor to larger clinical trials.

Ethical Considerations Patients participating in this trial will have suffered major intracranial haemorrhage with poor prospect of favourable neurological recovery even with maximal current treatment. In this situation, the potential benefits of the RT outweigh the foreseeable risks and on balance favour offering the study intervention to patients.

Patients enrolled in the study will receive additional computed tomography (CT) scans involving ionising radiation. These scans will exclude certain causes of haemorrhage (aneurysm) that would preclude safely administering the RT therapy. Diagnosis of aneurysm would however be of substantial benefit to the patient in determining their further clinical management. Volume STEALTH CT scans will be obtained prior to surgery and at 24-48 hours post-operatively to aid in navigating the RT catheter and to measure the degree of clot evacuation. To guide the number of passes of the RT catheter an on-table CT scan may be necessary intra-operatively. In total, the additional radiation dosage equates to approximately 4 milliSieverts (mSv), equivalent to approximately 1.5 years background radiation. Set against the potential benefits of RT this is not excessive.

Patients suitable for RT and fulfilling the inclusion and exclusion criteria, will, because of their condition, not be able to give informed consent. The nature of the pathology being studied means that a trial of a novel treatment cannot first be conducted in patients able to give their own consent. The investigators will approach family, relatives, and friends to discuss patients' expressed wishes towards participating in research and proceed with enrolment if the consultees are in agreement.

Objectives

* To determine the feasibility and efficacy of rheolytic thrombectomy for evacuating intraventricular haemorrhage, measured by computed tomography-based volumetric analysis
* To assess the safety of using RT in adult intraventricular haemorrhage

Study Design

Summary of Design Single centre prospective cohort study of 20 patients with IVH treated with RT

Study Centres

This is a single-centre study to be conducted at:

Addenbrooke's Hospital Cambridge University Hospitals NHS Foundation Trust Hills Road Cambridge CB2 0QQ

Sample Size Number of Participants 20 patients

Sample Size Determination From the investigators previous experience the sample size will be sufficient for a pilot study to evaluate the feasibility and safety of RT in IVH.

Study Duration Recruitment is expected to take up to 24 months.

Endpoints Primary Endpoint Clearance of intraventricular blood measured on computed tomography

Secondary Endpoints

* Presence of ependymal cells and/or neural tissue cells within effluent collected during operation
* 14-day survival
* Modified Rankin Score at 6 months
* Duration of External Ventricular Drainage
* Permanent CSF diversion (i.e. shunt)
* Intra- or post-operative rebleeding
* Culture-proven infection (meningitis/ventriculitis)

Study Participants Overall Description of Participants Adult patients admitted in coma with severe intraventricular haemorrhage requiring external ventricular drainage

Patient Withdrawal Patients or their nominated consultee are free to withdraw from the study at any time.

Patients will be withdrawn from the study following baseline CT angiography if an aneurysm is demonstrated that is thought to have possibly caused the IVH.

Patients withdrawn from the study prior to RT will be replaced to achieve to ensure a full assessment of feasibility and safety can be made.

Given the study involves a one-time intervention it is not envisaged patients will be withdrawn from follow-up after RT, unless requested by them or their nominated consultee.

Definition of the End of the Study The study will be terminated on completion of recruitment and 6-month follow-up of 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Coma at presentation (i.e. Glasgow Coma Score <9)
* At least 50% of lateral ventricles cast with blood
* Evidence of hydrocephalus or raised intracranial pressure and External Ventricular Drainage Indicated
* Surgery possible within 48 hours of ictus

Exclusion Criteria:

* Fixed and dilated pupils at presentation
* Uncorrectable coagulopathy or thrombocytopenia
* Aneurysm or arteriovenous malformation proven or suspected as the source of haemorrhage
* Large, predominant intracerebral haematoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Clearance of intraventricular blood measured on computed tomography | 96 hours

SECONDARY OUTCOMES:
14-day survival | 14 days
Modified Rankin Score at 6 months | 6 months
Duration of External Ventricular Drainage | 30 days
Permanent CSF diversion | 2 years
Intra- or post-operative rebleeding | 96 hours
Culture-proven CNS infection | 30 days